CLINICAL TRIAL: NCT03899467
Title: An Multi-Center, Randomized, Open-Label Study to Evaluate the Safety and Tolerability of GT0918 in Subjects With mHSPC and mCRPC Who Failed Either Abiraterone or Enzalutamide
Brief Title: The Safety and Tolerability of GT0918 in Subjects With mHSPC and mCRPC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Kintor Pharmaceutical Inc, (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GT0918-US-1002
Record Dates: First submitted 2019-03-27; First posted 2019-04-02 (Actual); Results first posted 2024-01-02 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Castrate Resistant Prostate Cancer (mCRPC); Metastatic Hormone-Sensitive Prostate Cancer (mHSPC)
MeSH Terms: interventions — proxalutamide; Androgen Receptor Antagonists

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: 400 mg /day of GT0918 (Experimental): Group 1: Post enzalutamide failure
  Group 2: Post abiraterone failure
  Interventions: Drug: GT0918
- Arm 2: 500 mg/day of GT0918 (Experimental): Group 1: Post enzalutamide failure
  Group 2: Post abiraterone failure
  Interventions: Drug: GT0918

INTERVENTIONS:
Drug: GT0918 — anti-tumor activity
  Other Names: proxalutamide; androgen receptor antagonist

SUMMARY:
This was a multiple-center, open-label, randomized, daily dose, two-sequence, expanded/phase II study in subjects with mHSPC or mCRPC who progressed after either abiraterone or enzalutamide treatment.

The objective of the study is to evaluate the safety and tolerability of proxalutamide and determine the RP2D for Ph III and/or other confirming studies.

Subjects will be randomized into the 2 treatment arms.

DETAILED DESCRIPTION:
This study is an open-label, randomized, expanded/phase II study in subjects with mHSPC or mCRPC who progressed after either abiraterone or enzalutamide. All subjects will be randomized to take 400 mg or 500 mg of GT0918 by oral administration once daily on an empty stomach (2-3 hours after a meal) for initial treatment of 6 months. Randomization of subjects will be stratified by prior therapy (abiraterone or enzalutamide).

Subjects will continue treatment with GT0918 (proxalutamide) at their assigned dose on an empty stomach until disease progression, intolerable toxicities (AEs), or withdrawn consent. A post-treatment period of 4 weeks will commence that concludes with an end-of-study visit.

Disease progression will be assessed by three methods over the duration of the study. Subjects will be assessed for biochemical (PSA) progression measured monthly, as well as radiographic progression by CT scan or/and bone progression by radionuclide bone scan every 12-weeks. Progressive disease will be considered on the occurrence of the first assessed progression event. Subjects with PSA progression only may continue the study until radiographic or bone progression at the discretion of the Investigator and with agreement by the sponsor or their authorized medical monitor.

ELIGIBILITY:
Inclusion criteria:

1. Signed informed consent obtained prior to any study-related procedure being performed.
2. Subjects at least 18 years of age or older at the time of consent.
3. Subjects with histologically confirmed mHSPC or mCRPC who received abiraterone or enzalutamide for the hormonal treatment of 6 months or longer.
4. Subjects with mHSPC are required to have no prior ADT (androgen deprivation therapy) or orchiectomy. For mCRPC, ongoing androgen deprivation therapy with a luteinizing hormonereleasing hormone (LHRH) "super-agonist" or antagonist, or bilateral orchiectomy. Serum testosterone level is < 50 ng/dL (< 0.5 ng/mL, < 1.7 nmol/L) at screening.
5. Metastatic disease documented by computed tomography (CT)/magnetic resonance imaging (MRI) or bone scan.
6. Progressive disease despite hormonal treatment with abiraterone or enzalutamide, but not both. However, if either of these 2 drugs was used less than 3 months due to toxicity, the patient is eligible. One line of chemotherapy is eligible. Progressive disease is defined by 1 or more of the following criteria:

   1. Subjects with a rising prostate specific antigen (PSA) value > 2 ng/mL in at least 2 measurements, at least 1 week apart. If the confirmatory PSA value is less than the screening PSA value, then an additional test for the rising PSA is required to document progression.
   2. Subjects with measurable disease, progression defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
   3. Subjects with metastatic bone disease, progression defined by 2 or more new lesions in a radionuclide bone scan.
7. ECOG performance status of 0-1
8. Screening blood counts of the following:

   1. Absolute neutrophil count ≥ 1500/μL
   2. Platelets ≥ 100,000/μL
   3. Hemoglobin > 9 g/dL (if asymptomatic).
9. Screening chemistry values of the following:

   1. Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 2.5 × upper limit of the normal reference range (ULN)
   2. Total bilirubin ≤ 2 × ULN
   3. Creatinine ≤ 1.5 × ULN
   4. Albumin > 2.8 g/dL.
10. At screening, life expectancy of at least 6 months.
11. Subjects whose partners are women of childbearing potential (WOCBP) must use an adequate method of birth control while on study drug and for at least 3 months after discontinuation of study drug.
12. Subject is willing and able to comply with all protocol required visits and assessments.

Exclusion criteria:

1. Discontinuation of enzalutamide or abiraterone less than 3 weeks prior to the start of study medication.
2. Prior chemotherapy and experimental therapy (Poly (ADP-ribose) polymerase (PARP) or checkpoint inhibitor)
3. Ongoing acute treatment-related toxicity associated with a previous therapy greater than grade 1 except for grade 2 alopecia or neuropathy.
4. History of impaired adrenal gland function (e.g., Addison's disease, Cushing's syndrome).
5. Known gastrointestinal disease or condition that affects the absorption of proxalutamide.
6. History of congestive heart failure New York Heart Association (NYHA) class III or IV or uncontrolled hypertension at screening.
7. History or family history of long QT syndrome, or ECG corrected QT interval equal to and over 500 ms (CTCAE grade 2) at baseline.
8. History of other malignancy within the previous 3 years, except basal cell or squamous cell carcinoma, or non-muscle invasive bladder cancer.
9. Use of systemic glucocorticoid (e.g., prednisone, dexamethasone) within 14 days prior to the start of study medication. Inhaled or topical steroids are allowed.
10. Co-administration of CYP3A4 ligands that serve as substrates or induce or inhibit the enzyme.
11. Prior use of any herbal products known to decrease PSA levels (e.g., PC-SPES or saw palmetto) within 30 days prior to the start of study medication.
12. Major surgery within 30 days prior to the start of study medication.
13. Blood transfusion (including blood products) within 1 week of screening.
14. Serious persistent infection within 14 days prior to the start of study medication.
15. Serious concurrent medical condition including CNS disorders.
16. Previous history of difficulty swallowing capsules.
17. Known hypersensitivity to GT0918 or its excipients.
18. Any condition that, in the opinion of the investigator, would impair the subject's ability to comply with study procedures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-09-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University Cancer & Blood Center, Athens, Georgia
  - Norton Cancer Institute, Louisville, Kentucky
  - Chesapeake Urology Research Associates, Towson, Maryland
  - G U Research Network, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New York Cancer & Blood Specialists, East Setauket, New York
  - New York Cancer & Blood Specialists, The Bronx, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - Greenville Health System, Greenville, South Carolina
  - Mary Crowley Cancer Research, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The anticipated 60 subjects would be enrolled per protocol; Actually, total 61 subjects were randomized to take 400 mg or 500 mg of GT0918.
Pre-assignment Details: The anticipated 60 subjects would be enrolled per protocol; Actually, total 61 subjects were randomized to take 400 mg or 500 mg of GT0918; 31patients were enrolled in 400mg arm and 30 patiens were enrolled in 500mg arm respectively. Randomization of subjects were stratified by prior therapy (abiraterone or enzalutamide).The post enzalutamide and post abiraterone groups were not pre-specified to be analyzed and as separate Arms/Groups.
Groups:
- Arm 1: 400 mg /Day of GT0918; Arm 2: 500 mg/Day of GT0918: Group 1: Post enzalutamide failure
  Group 2: Post abiraterone failure
  GT0918: anti-tumor activity
Period: Overall Study
Arm/Group | Arm 1: 400 mg /Day of GT0918 | Arm 2: 500 mg/Day of GT0918
Started | 31 | 30
Completed | 19 | 22
Not Completed | 12 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: 400 mg /Day of GT0918 | Arm 2: 500 mg/Day of GT0918 | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.8 (8.71) | 74.3 (7.39) | 73.5 (8.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 31 | 30 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 27 | 29 | 56
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 7 | 9
  White | 27 | 22 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
BMI [Median (Full Range); unit: Kg/mg^2] | 29.4 [17.7 to 41.2] | 29.1 [22.6 to 42.9] | 29.3 [17.7 to 42.9]

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Safety and Tolerability of GT0918 and Select the RP2D for Future Clinical Trial Study.
Description: To evaluate the safety and tolerability of GT0918 assessed by AEs, SAEs between 400 mg arm vs. 500 mg arm with mHSPC or mCRPC who failed either abiraterone or enzalutamide treatment The percetage of AE and SAE would be evaluated in subjects with mHSPC and to determine the recommended Phase II dose (RP2D) over 6 months or longer treatment
Time Frame: Average of 24 weeks, up to a maximum of 30 weeks
Population: The Safety Analysis Set (SS) included all 61 subjects who have taken at least one dose of study medication;31 subjects and 30 subjects were incuded in 400mg daily arm and 500mg daily arm,respevtively
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: 400 mg /Day of GT0918 | Arm 2: 500 mg/Day of GT0918
Number analyzed (Participants) | 31 | 30
Participants
  TEAE | 28 | 29
  SAE | 6 | 12

2. Secondary Outcome: The Percentage of Subjects Achieving a ≥50% Reduction in PSA at 12 Weeks and 24 Weeks
Description: The percentage of subjects achieving a ≥50% reduction in PSA at 3 months (12 weeks) as compared to baseline (study entry) was determined.
Time Frame: 24 weeks
Population: The Full Analysis Set (FAS) will include subjects who have post-baseline PSA assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: 400 mg /Day of GT0918 | Arm 2: 500 mg/Day of GT0918
Number analyzed (Participants) | 22 | 18
Participants
  PSA ≥50% reduction at Week 12 | 2 | 1
  PSA ≥50% reduction at Week 24 | 1 | 1

3. Secondary Outcome: Time to PSA Progression
Description: Time to PSA Progression in 400mg group and 500mg group
Time Frame: 24 weeks
Population: The Full Analysis Set (FAS) will include subjects who have at least one post-treatment tumor assessment.
Measure: Median (Full Range); unit: day
Arm/Group | Arm 1: 400 mg /Day of GT0918 | Arm 2: 500 mg/Day of GT0918
Number analyzed (Participants) | 22 | 18
day | 85 [29 to 168] | 83.5 [27 to 168]

4. Secondary Outcome: PSA Maximum Change at 12 Weeks
Description: The percentage of change of PSA from baseline at Week 12 was calculated. Maximum percentage change of PSA from baseline at any time was calculated.
Time Frame: 24 weeks
Population: The percentage change of PSA from baseline at any visit was calculated for the FAS
Measure: Median (Full Range); unit: percent change
Groups:
- GT0918 400mg Daily; GT0918 500mg Daily: Group 1: Post enzalutamide failure
  Group 2: Post abiraterone failure
  GT0918: anti-tumor activity
Arm/Group | GT0918 400mg Daily | GT0918 500mg Daily
Number analyzed (Participants) | 29 | 29
percent change | -5.58 [-99.1 to 25948.6] | 45.61 [-97.3 to 470.3]

ADVERSE EVENTS:
Time Frame: Average of 24 weeks, up to a maximum of 30 weeks
Description: An adverse event (AE) is any symptom, physical sign, syndrome, or disease that either emerges or, if present at screening, worsens during the study, regardless of the suspected cause of the event.The period of collection of AEs is from the time of first dose to the last dose of study drug or EOS visit. The 30-day safety follow up "window" is set to capture possibly drug-related AE and/or SAE.
Arm/Group | Arm 1: 400 mg /Day of GT0918 | Arm 2: 500 mg/Day of GT0918
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 6/31 | 12/30
Other Adverse Events (participants affected / at risk) | 28/31 | 26/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: 400 mg /Day of GT0918 (N=31) | Arm 2: 500 mg/Day of GT0918 (N=30)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Dry gangrene (Vascular disorders) | 1 (1) | 0 (0)
COVID-19 pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: 400 mg /Day of GT0918 (N=31) | Arm 2: 500 mg/Day of GT0918 (N=30)
Constipation (Gastrointestinal disorders) | 11 (11) | 13 (13)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4)
Nausea (Gastrointestinal disorders) | 8 (8) | 7 (7)
Fatigue (General disorders) | 15 (15) | 16 (16)
Asthenia (General disorders) | 1 (1) | 4 (4)
Oedema peripheral (General disorders) | 8 (8) | 7 (7)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 7 (7)
Weight decreased (Investigations) | 5 (5) | 10 (10)
Decreased appetite (Metabolism and nutrition disorders) | 9 (9) | 14 (14)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2)
Dysgeusia (Nervous system disorders) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 3 (3)
Depression (Psychiatric disorders) | 4 (4) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3)
Gait disturbance (General disorders) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Hypersomnia (Nervous system disorders) | 2 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 2 (2) | 1 (1)
Confusional state (Psychiatric disorders) | 3 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT03899467/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT03899467/ICF_001.pdf